CLINICAL TRIAL: NCT03534609
Title: Exploratory Evaluation of the Lutronic Genius System for Treatment of the Neck
Brief Title: Lutronic Genius System for Neck Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CynosureLutronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L18000
Record Dates: First submitted 2018-04-16; First posted 2018-05-23 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Wrinkle; Skin Laxity; Skin Texture Disorder
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Genius System Neck Treatment (Experimental): Lutronic Genius System treatment of lines, wrinkles, and texture concerns on the neck.
  Interventions: Device: Lutronic Genius System

INTERVENTIONS:
Device: Lutronic Genius System — Treatment of the neck using the Lutronic Genius System

SUMMARY:
The Genius system is substantially equivalent to the Infini device (K121481). The study is a prospective, multi-site, non-randomized study of up to 30 treated subjects presenting for treatment of mild to moderate lines, wrinkles, textural concerns, and/or skin laxity of the neck.

DETAILED DESCRIPTION:
At enrollment, standardized baseline/pretreatment 2D and 3D images will be obtained from each subject. Study subjects will receive three neck treatments completed 30 days apart. Subjects will be contacted via a phone call 3 days following each treatment to assess for adverse events and expected treatment effects. Effectiveness assessments will occur prior to Treatments #2 and #3, and a follow-up visit will be completed at 90 days following Treatment #3. Each assessment visit will include efficacy, adverse events, and expected treatment effects assessments, and post-treatment 2D and 3D digital images will be captured.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years and older.
2. Subject in good health.
3. Fitzpatrick Skin Type I to VI.
4. Mild to moderate lines, wrinkles, textural concerns, and/or skin laxity of the neck.
5. Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
6. Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
7. Post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study.
8. Absence of physical or psychological conditions unacceptable to the investigator.
9. Willingness and ability to provide written consent for study-required photography and adherence to photography procedures (i.e., removal of jewelry and makeup).
10. Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.

Exclusion Criteria:

1. Presence of an active skin condition or infection in the treatment area such as sores, Psoriasis, eczema, rash, severe active inflammatory acne or oral herpes simplex breakout.
2. History of skin disorders, keloid scarring, and/or abnormal wound healing.
3. Open wounds or lesions in the area(s) to be treated.
4. Inability to understand the protocol or to give informed consent.
5. History of chronic drug or alcohol abuse.
6. History of vascular disease.
7. History of bleeding disorders.
8. BMI equal to or greater than 30.
9. Subjects who are pregnant, nursing, or anticipate a pregnancy during the length of the trial.
10. Subjects with current skin cancer or other malignant disease including pre-malignant moles.
11. Poorly controlled medical condition that could compromise wound healing or increase risk of infection such as an impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications, radiation therapy, or chemotherapy.
12. Subjects with implanted medical devices: pacemaker, cardioverts, superficial metal within the treatment area, and other implantable devices or synthetic fillers.
13. Subjects with sensitivity or allergy to gold.
14. Subjects with sensitivity or allergy to local anesthetics such as lidocaine or tetracaine.
15. Concurrent enrollment in any study involving the use of investigational devices or drugs.
16. History of surgical or cosmetic treatments in the area(s) to be treated within the past six months.
17. History or current use of the following prescription medications:

    1. Daily anticoagulants, aspirin, iron supplements, herbal supplements such as ginkgo, ginseng or garlic within the past two weeks;
    2. Topical retinoid within the past one week; and
    3. Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Masked qualitative assessment of improvement | From baseline to 90 days following the last treatment
  An assessment of paired pre- and post-treatment photographs will be conducted by blinded assessors evaluating for improvement in neck appearance from pre- to post-treatment. The assessors choose the photo they believe to be the post-treatment photo, i.e., Left photo or Right photo.

SECONDARY OUTCOMES:
Clinician aesthetic improvement | From baseline to Days 90 following the last study treatment.
  Overall aesthetic improvement based on completion of the Clinician Global Aesthetic Improvement Scale, a 5-point scale (0-4) that rates global aesthetic improvement from the pre-treatment appearance with 4 being 'Very Much Improved' and 0 being 'Worse'. The scale will be administered based on a live assessment of the subject while referring to the subject's pre-treatment photographs, and based on a comparison of the subject's pre-treatment photographs to the Day 90 follow-up photographs.
Subject aesthetic improvement | From baseline to Days 90 following the last study treatment.
  Overall aesthetic improvement based on completion of the Subject Global Aesthetic Improvement Scale, a 5-point scale (0-4) that rates global aesthetic improvement from the pre-treatment appearance with 4 being 'Very Much Improved' and 0 being 'Worse'. Subjects will complete the scale based on a live assessment while referring to a hand mirror and their pre-treatment photographs, and based on a comparison of their pre-treatment photographs to their Day 90 follow-up photographs.
Patient Satisfaction | From baseline to 90 days following the last study treatment
  Patient satisfaction will be evaluated based on subjects' completion of a patient satisfaction questionnaire while referring to a hand mirror and their pre-treatment and their Day 90 follow-up photographs.
Treatment-related pain | For the duration of each study treatment which typically can last up to approximately 90 minutes.
  During each study treatment, subjects' pain levels will be monitored using a validated Numeric Rating Scale (0-10), with 0 being 'No Pain' and 10 being 'Worse Possible Pain'.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Larson, MBA, Study Director — Sponsor GmbH
Locations (1):
- Laser and Skin Surgery Center of New York, New York, New York, United States